CLINICAL TRIAL: NCT06103227
Title: The Effect of Low Doses of Intermediate Acting Corticosteroids on the Prolongation of Pregnancy in Threatened Preterm Birth
Brief Title: The Effect of Low Doses of Prednisone on the Prolongation of Pregnancy in Threatened Preterm Birth
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Mostar (Other)
Responsible Party: Principal Investigator, Nikolina Penava, Maternal-fetal medicine specialist, University of Mostar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1236/23
Record Dates: First submitted 2023-10-21; First posted 2023-10-26 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Preterm Birth
Keywords: Premature birth, sterile inflammation, prednisone
MeSH Terms: conditions — Premature Birth | interventions — Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low dose of prednisone group (Experimental): Low-dose prednisone was used for a total of three weeks from the initiation of RDS prophylaxis, following two-day tocolysis and magnesium sulphate for neuroprotection.
  Interventions: Drug: Prednisone 5Mg
- Standard therapy group (Active Comparator): Two-day tocolysis and RDS prophylaxis, plus neuroprotection with magnesium sulphate.
  Interventions: Drug: Prednisone 5Mg

INTERVENTIONS:
Drug: Prednisone 5Mg — Prednisone administered for three weeks. If pregnant women weighs less than 90 kg , she will receive prednisone on altering days instead of every morning for pregnant women weighing more than 90 kg.

SUMMARY:
The goal of this clinical trial is to test the effect of a low dose of prednisone in the prevention of preterm labour in singleton pregnancies. The main question it aims to answer is whether prednisone prolongs singleton pregnancy in threatened preterm birth and reduces mortality and morbidity of newborns without harmful consequences for the mother and the foetus. Participants will be:

* administered low dose of prednisone in a period of a total of 3 weeks on top of standard therapy
* drown blood for standard laboratory tests
* cervical swab and urine for urine culture will be taken, and
* asked to sign Informed Consent The researcher will compare a low dose of prednisone to standard therapy.

DETAILED DESCRIPTION:
Prematurity is the leading cause of infant mortality and is associated with an increased risk of respiratory, neurological and metabolic disorders in survivors. Approximately 15 million babies are born preterm annually worldwide. Despite the rapid development of pharmacotherapy, there was no significant decline in premature birth (PTB) rates. So far, the most useful intervention for improving neonatal outcomes in premature children has been the antenatal administration of long-acting corticosteroids (CSs). Although the underlying causes of PTB are numerous, it is well established that infection and inflammation represent a highly significant risk factor for spontaneous PTB, characterized by the significant production of inflammatory mediators that lead to the weakening of the foetal membranes, cervical stroma and contraction of the myometrium. There is increasing evidence of the presence of sterile inflammation (intra-amniotic inflammation without the presence of microorganisms) in PTB with both intact membranes and preterm premature rupture of membranes (PPROM). CS and non-steroidal anti-inflammatory drugs (NSAID) are used today to treat most inflammatory diseases. NSAIDs are used as tocolytics. Indomethacin, one of the most commonly used NSAID tocolytics, has been associated with oligohydramnios and premature closure of the foetal ductus arteriosus when used for prolonged periods. As far back as 1972, Liggins and Howie proved that antenatal administration of CS reduces the incidence and severity of respiratory distress syndrome (RDS) and mortality of premature infants. Meta-analyses have confirmed a lower rate of intraventricular haemorrhage and necrotic enterocolitis in premature infants whose mothers received RDS prophylaxis. Therefore, their application proved to be the most useful intervention for improving neonatal outcomes in threatening PTB. Today, CS is a part of standard therapy for treating systemic autoimmune diseases and acts as a suppressor of immune response. Long acting CSs cross the placental barrier and are used to treat the foetus (foetal lupus, congenital adrenal hyperplasia, prevention of respiratory distress syndrome), and intermediate acting drugs are used to treat maternal diseases as they have a low affinity for passing through the placenta. The effect of low doses of intermediate acting corticosteroids on the prolongation of pregnancy in threatened preterm birth has not yet been studied. Given that PTB is a syndrome characterized by a strong inflammatory response, we present the hypothesis that low doses of an intermediate acting CS for 3 weeks after tocolysis and RDS prophylaxis help prolong singleton pregnancy in women with threatening PTB, without harmful consequences for mother and child.

ELIGIBILITY:
Inclusion Criteria:

- primiparity, singleton pregnancy between 24+0 and 34+0 weeks, and signs of threatened PTB at admission. Threatened PTB was defined as regular uterine contractions (>4 in 20 minutes or >8 in 60 minutes), with or without bleeding, along with cervical dilation greater than 2 cm or cervical length less than 20 mm, confirmed by transvaginal ultrasound or clinical progression.

Exclusion Criteria:

- contraindications to tocolysis or systemic corticosteroid (CS) therapy, such as intrauterine fetal death, lethal fetal anomaly, abnormal CTG recording, severe preeclampsia or eclampsia, hemodynamically significant bleeding, infection, uncontrolled diabetes, ongoing CS therapy for underlying conditions, severe liver impairment, or preterm prelabour rupture of membranes.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 26 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Number of days by which singleton pregnancies with threatened preterm birth are prolonged | 10 weeks (from 24th till 34th week of pregnancy)
  Prolongation of singleton pregnancy in threatened preterm birth

SECONDARY OUTCOMES:
Change of mortality and morbidity | 10 weeks (from 24th till 34th week of pregnancy)
  Change mortality and morbidity of newborns without harmful consequences for the mother and the foetus.

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinical Hospital, Mostar, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: No